CLINICAL TRIAL: NCT04984967
Title: Comparison of Two Techniques of Peripheral Venous Catheterization in Newborns : Insertion on Micro-guide Versus Conventional Insertion, Without Micro-guide
Brief Title: Interest of Peripheral Venous Catheter Insertion Using a Micro-guide in Neonatology
Acronym: EASYCATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RECHMPL20_0410
Record Dates: First submitted 2021-06-03; First posted 2021-08-02 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Newborns; Neonatology; Intensive Care
Keywords: Newborn infant; Intensive care; vascular access; Peripheral intravenous catheterization

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Peripheral venous catheterization is perform by a nurse. The placement characteristics are evaluated by the investigator, blind of the condition of placement if possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insertion of peripheral venous catheter with micro-guide (Experimental)
  Interventions: Device: Insertion of peripheral venous catheter with micro-guide
- Classic insertion of peripheral venous catheter, without micro-guide (Other)
  Interventions: Other: Classic insertion of peripheral venous catheter, without micro-guide

INTERVENTIONS:
Device: Insertion of peripheral venous catheter with micro-guide — After antisepsis, the vein is punctured using a needle. Then the micro-guide is inserted to the first landmark, which indicates the passage of the micro-guide beyond the end of the needle. After the needle removed, the peripheral venous catheter is placed on the micro-guide. The guide is then removed, the peripheral venous catheter can be used.
  Arms: Insertion of peripheral venous catheter with micro-guide
Other: Classic insertion of peripheral venous catheter, without micro-guide — After antisepsis, the catheter is introduced into the vein by a needle which is subsequently removed while the catheter remains in place.
  Arms: Classic insertion of peripheral venous catheter, without micro-guide

SUMMARY:
Peripheral venous catheterization represents the preferential option for term or preterm infant care in order to start drug treatment or hydration, or perform anesthesia.

However, the peripheral venous access is associated in approximately 50% of cases with a failure of the insertion on the first attempt in an emergency context. Using a micro-guide may facilitate the peripheral venous catheterization in newborns, by guiding the catheter in the vein and, thereby reduce the risk of transfixion of the vascular lumen.

ELIGIBILITY:
Inclusion Criteria:

* Newborn admitted in the department of neonatal medicine and pediatric intensive care, at Montpellier University Hospital

Exclusion Criteria:

* Term neonate > 28 days
* Premature neonate > 41 weeks of corrected gestational age
* Exclusive requirement for an umbilical venous catheter, in the context of neonatal resuscitation
* Exclusive requirement for an epicutaneous-cava catheter, in the context of prolonged parenteral nutrition.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Success of peripheral venous catheterization at the first attempt | Up to 5 minutes after the success of the placement
  The success of the placement is defined by the arrival of blood in the transparent chamber downstream of the needle during the placement, and by the absence of painful reaction and edema near the insertion site, indicating extravasation or extravascular passage, after flushing the catheter with 0.5 to 1 ml of isotonic saline. The success will be confirmed by retesting flush after securing the peripheral venous catheter in a dressing, within 3 to 5 minutes of successful puncture.

SECONDARY OUTCOMES:
Efficiency of the technique | Up to 4 days.
  Assessed by the number of venipuncture attempts.
Efficiency of the technique | Up to 4 days.
  Assessed by the duration of the installation (time from the end of skin asepsis to the end of the occlusive dressing).
Efficiency of the technique | Up to 4 days.
  Assessed by the requirement to insert a central venous line directly linked to failure of peripheral venous catheterization.
Efficiency of the technique | Up to 4 days.
  Assessed by the reason for removal of peripheral venous catheter (ie, elective removal or removal for the occurrence of adverse events, see below).
Adverse events | Up to 4 days.
  Specifically associated with the micro-guide: section, intravascular migration, venous transfixion.
Adverse events | Up to 1 month.
  Common to the placement of any peripheral venous catheter, regardless of the insertion technique : puncture of an artery, pain, hemorrhage at the puncture site, phlebitis, thrombosis, infection, obstruction and subcutaneous diffusion of the infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Montpellier, Montpellier, France